CLINICAL TRIAL: NCT04971213
Title: HIgh Flow Nasal Cannula Versus Noninvasive Ventilation for Acute Cardiogenic PuLmonary Oedema With Acute Respiratory Failure in an ED
Brief Title: HIgh Flow Versus NIV for Acute Cardiogenic PuLmonary Oedema With Acute Respiratory Failure in an ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIPPOLYTE
Record Dates: First submitted 2021-07-06; First posted 2021-07-21 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Cardiogenic Pulmonary Edema
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non Invasive Ventilation (Active Comparator): Bilevel non-invasive ventilation. Support pressure will be set to obtain a 6-8 mL/kg of predicted body weight PEEP will be set within 5-10 cmH2O and FiO2 for a SpO2 equal or over 94% target. (92% in patients with chronic respiratory failure) All settings will be adjusted according tolerance of the patient.
  Interventions: Device: Non invasive ventilation
- High-flow nasal cannula heated and humidified oxygen (Experimental): Flow will be set at 60 L/min and ajusted according the tolerance of the patient.
  FiO2 will be set according a SpO2 equal or over 94% target. (92% in patients with chronic respiratory failure)
  Interventions: Device: High-flow nasal cannula heated and humidified oxygen

INTERVENTIONS:
Device: Non invasive ventilation — Emergency and transport ventilator (Monnal T60, Airliquide, Antony, France)
  Arms: Non Invasive Ventilation
Device: High-flow nasal cannula heated and humidified oxygen — AirVO2 device (Fisher and Paykel, New Zealand)
  Arms: High-flow nasal cannula heated and humidified oxygen

SUMMARY:
The purpose of this study is to compare non invasive ventilation to high flow nasal cannula oxygen for the management of patients admitted with an acute respiratory failure due to an acute cardiogenic pulmonary edema.

DETAILED DESCRIPTION:
Acute cardiogenic pulmonary oedema is a leading cause of acute respiratory distress in patients admitted in an Emergency Department. With diuretics and nitrite derivative, noninvasive ventilation is the first-line treatment of acute pulmonary oedema recommended by the European Society of Cardiology. Noninvasive ventilation is able to reduce the respiratory rate faster than standard oxygen therapy, to improve oxygenation, and some data suggest it could reduce the mortality rate. NIV may be poorly tolerated in certain patients, in whom it is associated with failure of treatment and poor outcomes. High-flow nasal cannula heated and humidified oxygen (HFNO) is a ventilatory support used in ICU and recently introduced in Emergency Departments. As compared NIV and standard oxygen therapy, HFNO reduces the mortality rate in patients with acute hypoxemic respiratory failure hospitalized in an ICU. In addition, in these patients, HFNO is also better tolerated than noninvasive ventilation. Some data suggested HFNO is superior to standard oxygen therapy in acute pulmonary oedema and could have a similar clinical effect to NIV. However, there is no research that has compared tolerance of patients admitted in an ED with acute pulmonary oedema and treated by HFNO or NIV.

Included patients will be treated with NIV or HFNO. NIV will be provided with an emergency and transport ventilator (Monnal T60, Airliquide, Antony, France) and HFNO will be provided with an AirVO2 device (Fisher and Paykel, New Zealand). Patients will be treated in an Emergency Department immediately after their admission and their consent. Treatment will be provided for a minimum of one hour. Tolerance of patients will be measured under treatment using a comfort numerical scale from 0 - well comfortable to 10 extremely uncomfortable. Clinical and biological patterns will be also recorded. Patients will be followed from their inclusion to 28 days after their inclusion.

ELIGIBILITY:
Inclusion Criteria:

* age over or equal 18 years old
* admitted in an Emergency Department
* acute respiratory failure defined by a respiratory rate over or equal 25 breathes/min or signs of increased work of breathing
* clinical suspicion of acute heart failure defined bu the European Cardiologic Society.

Exclusion Criteria:

* patient requiring immediate invasive mechanical ventilation
* neurologic distress defined by a Glasgow Coma Scale under 13
* haemodynamic failure defined by a Mean Blood Pressure under 65 mmHg or patient requiring catecholamines

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Respiratory rate | 60 minutes
  Evolution of the respiratory rate within 60 minutes following the beginning of the treatment

SECONDARY OUTCOMES:
Clinical paterns | 15, 30, 60, 90 minutes after the treatment's beginning
  Respiratory rate in breaths/min, heart rate (beats/min), arterial blood pressure (mmHg), signs of increased work of breathing
Arterial blood gas | 1 hour after the treatment beginning
  PaCO2 (mmHg), PaO2 (mmHg), pH
Proportion of patients dying | 28 days
  Patient dying within 28 days
Proportion of patients requiring invasive mechanical ventilation | 28 days
  Mechanical ventilation within 28 days.
Comfort of patient according a numerical scale from 0 to 10 | 30, 60 minutes after the treatment's beginning
  Comfort will be assessed using a numerical scale.
Evolution of dyspnea according a Modified Borg Scale | 15, 30, 60, 90 minutes after the treatment's beginning
  Dyspnea score will be recorded by the patient using a Modified Borg scale for dyspnea
ROX index | 15, 30, 60, 90 minutes after the treatment's beginning
  Rox Index was measured as following : (SpO2/FiO2)/RR
Proportion of patients responding to the ventilatory support | 15, 30, 60, 90 minutes after the treatment's beginning
  Patients with a respiratory rate under or equal to 25 AND without signs of increased work of breathing.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin ALOS, MD, Study Chair — CHU Poitiers; Nicolas MARJANOVIC, MD PhD, Principal Investigator — CHU Poitiers; Jérémy Guenezan, MD, Study Chair — CH Nord-Vienne; Maxime Jonchier, MD, Study Chair — CHU de Poitiers (Site de Montmorillon)
Locations (1):
- CHU Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marjanovic N, Piton M, Lamarre J, Alleyrat C, Couvreur R, Guenezan J, Mimoz O, Frat JP. High-flow nasal cannula oxygen versus noninvasive ventilation for the management of acute cardiogenic pulmonary edema: a randomized controlled pilot study. Eur J Emerg Med. 2024 Aug 1;31(4):267-275. doi: 10.1097/MEJ.0000000000001128. Epub 2024 Feb 16. PMID 38364020